CLINICAL TRIAL: NCT03791060
Title: An Open-label Proof of Concept Study Regarding the Use of Secukinumab (Cosentyx) in Patients With Necrobiosis Lipoidica Diabeticorum (NLD)
Brief Title: Secukinumab for NLD (Cosentyx) in Patients With Necrobiosis Lipoidica Diabeticorum (NLD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely due COVID-19 pandemic and did not resume; participants are no longer being examined or receiving intervention.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Martina Porter, Assistant Professor of Dermatology, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P000634
Record Dates: First submitted 2018-12-21; First posted 2019-01-02 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Necrobiosis Lipoidica Diabeticorum
Keywords: Necrobiosis lipoidica; NLD
MeSH Terms: conditions — Necrobiosis Lipoidica | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Secukinumab Subcutaneous Injection (Experimental): 300 mg q weekly for 5 weeks followed by 300 mg q 4 weeks.
  Each subject will receive 300mg of Secukinumab by using 2 syringes of 150mg each as a subcutaneous injection at weeks 0,1,2,3,4 then every 4 weeks for a total of 9 doses over 24 weeks.
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — Secukinumab is selective for human IL-17A and potently neutralizes the bioactivity of this cytokine. IL-17A is the central cytokine in multiple autoimmune and inflammatory processes. It is being recognized as one of the principal pro-inflammatory cytokines in autoimmune diseases such as psoriasis, PsA and AS, uveitis and is thought to play a role in other inflammatory conditions.
  Other Names: cosentyx

SUMMARY:
This study investigates the efficacy of secukinumab in necrobiosis lipoidica diabeticorum (NLD).

DETAILED DESCRIPTION:
Necrobiosis lipoidica diabeticorum (NLD) is a rare granulomatous condition of the skin often presenting with papules and eventually atrophic plaques, most commonly on the distal extensor lower extremities, which can be painful and disfiguring. Currently no FDA-approved treatment exists, and no well-established treatment algorithm has been described. Reports on successful therapeutic interventions have generally been small and inconsistent.

Recent literature expanding on the previously poorly understood pathogenesis of NLD has suggested a potential role for IL-17 in the development of this condition. Thus blockade of IL-17 may be a potential therapeutic strategy in patients with NLD. Secukinumab (Cosentyx) is a human monoclonal antibody that targets IL-17a and is FDA approved for the treatment of psoriasis.

This open-label, proof of concept study regarding the use of Secukinumab in patients with NLD may be a first step in elucidating and defining a treatment for this chronic and potentially debilitating condition for which no FDA approved treatment currently exists.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18 and over
* Previous diagnosis of biopsy-proven NLD
* Active NLD lesions, defined as

  * clinical signs of inflammation, for example erythematous margins, sensations of itch, pain, dysaesthesia
  * lesions increasing in size or appearance of new lesions within the last 3 months
  * ulcerations
* Subjects must be able to understand and communicate with the investigator and comply with the requirements of the study and must give a written, signed and dated informed consent before any study related activity is performed.

Exclusion Criteria:

* History of an ongoing, chronic or recurrent infectious disease, or evidence of tuberculosis infection as defined by a positive QuantiFERON TB-Gold test at screening.
* Are currently pregnant, breastfeeding, or planning to get pregnant during the study.
* Previous hypersensitivity reaction to secukinumab or to any of the components.
* History of Inflammatory Bowel Disease (Crohn's Disease or Ulcerative Colitis)
* Allergy to Latex
* Currently on any other immunosuppressant systemic medication or within 28 days of baseline visit
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unwilling to use effective contraception during the study and for 16 weeks after stopping treatment.
* Subjects with a serum creatinine level exceeding 176.8 μmol/L (2.0 mg/dL)
* Screening total WBC count <2,500/μL, or platelets <100,000/μL or neutrophils <1,500/μL or hemoglobin <8.5 g/dL
* Known infection with HIV, hepatitis B or hepatitis C at screening or randomization. Patients who are Hepatitis B Core antibody and/or Hep B Surface Antigen positive will be excluded from this study. Patients who are Hepatitis C ab positive will also be excluded from this study.
* History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years (except for non-melanoma skin cancer and carcinoma in situ of the cervix)
* Are participating in another study using an investigational agent or procedure during participation in this study or within 28 days prior to baseline visit.
* Plans for administration of live vaccines during the study period or 6 weeks prior to randomization
* Any other procedural treatment for NLD with 28 days prior to baseline visit, including phototherapy, surgical intervention, laser therapy, or cryotherapy.
* Any other active skin disease or condition (e.g., bacterial, fungal or viral infection) that may interfere with assessment of NLD;
* Underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal) which in the opinion of the investigator significantly immunocompromises the subject and/or places the subject at unacceptable risk for receiving an immunomodulatory therapy

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2021-01-17 (Actual); Study Completion 2021-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexa Kimball, MD MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No screenfailures for the study
Groups:
- Secukinumab Subcutaneous Injection: 300 mg q weekly for 5 weeks followed by 300 mg q 4 weeks.
  Each subject will receive 300mg of Secukinumab by using 2 syringes of 150mg each as a subcutaneous injection at weeks 0,1,2,3,4 then every 4 weeks for a total of 9 doses over 24 weeks.
  Secukinumab: Secukinumab is selective for human IL-17A and potently neutralizes the bioactivity of this cytokine. IL-17A is the central cytokine in multiple autoimmune and inflammatory processes. It is being recognized as one of the principal pro-inflammatory cytokines in autoimmune diseases such as psoriasis, PsA and AS, uveitis and is thought to play a role in other inflammatory conditions.
Period: Overall Study
Arm/Group | Secukinumab Subcutaneous Injection
Started | 4
Completed | 3
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Patient characteristics and demographic data will be presented using descriptive statistics.
Arm/Group | Secukinumab Subcutaneous Injection
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Family history of diabetes [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Score of Participants Who Received Investigator Global Assessment Scores
Description: Number of patients who received Investigator Global Assessment Scores rating their remission or clinical improvement as measured at week 24.
  The minimum score is zero and the maximum score is 6. A larger score is worse. Score Descriptions:
  0. Completely clear: except for possible residual hyperpigmentation
  1. Almost clear: very significant clearance (about 90%); however, patchy remnants of dusky erythema and/or very small ulcerations
  2. Marked improvement: significant improvement (about 75%); however, a small amount of disease remaining (i.e. remaining ulcers, although have decreased in size, minimal erythema and/or active boarder)
  3. Moderate improvement: intermediate between slight and marked; representing about 50% improvement
  4. Slight improvement: some improvement (about 25%); however, significant disease remaining (i.e. remaining ulcers with only minor decrease in size, erythema or boarder activity)
  5. No change from baseline
  6. Worse
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Secukinumab Subcutaneous Injection
Number analyzed (Participants) | 4
score on a scale | 4 (0.81)

2. Secondary Outcome: Histology
Description: Number of subjects achieving improvement based upon histological score. The score is calculated by adding subscores as listed below, which will be evaluated by the dermatopathologist. Average of pre and post scores and overall change in score will be calculated and compared using a paired T-test.
  1. Inflammatory infiltrate (0, none; 1, slight; 2, moderate; 3, severe)
  2. collagen degeneration (0, none; 1, slight; 2, moderate; 3, severe)
  3. epithelioid histiocytes, (0, none; 1, slight; 2, moderate; 3, severe)
  4. qualitative expression of IL-17 (0, none; 1, slight; 2 moderate; 3, severe)
  Histologic analysis not performed as study was terminated prematurely.
Time Frame: 26 weeks
Population: Histologic analysis was not performed on any subjects. Study was terminated prematurely and performing histology analysis for 4 subjects would not have reflected appropriate results. Dermatopathologist didnt evaluate biopsies, only confirm diagnosis for eligibility.
Arm/Group | Secukinumab Subcutaneous Injection
Number analyzed (Participants) | 0

3. Secondary Outcome: Pain Score Baseline and Week 24
Description: Number of patients who completed the self-reported pain and stinging intensity during and directly after treatment with Secukinumab injections
  A Pain Score will be calculated based upon the Wong-Baker Faces Pain rating Scale (10-point pain score), which has been widely used to rate pain in both children and adults and has also been used in dermatology clinical trials.
  Scale score 0-10, higher score means worse outcome:
  0 = No hurt 2 = Hurts a little bit 4 = Hurts a little bit more 6 = Hurts even more 8 = Hurts whole lot 10 = Hurts worst Response based on an improvement from baseline in the Wong-Baker pain score at all scheduled time points will be calculated. We will compare pre and post treatment pain values and categorize patients as (i) Resolved (ii) Improved (iii) Stable (iv) Worsened
Time Frame: Baseline and Week 24
Population: Analyzed mean scores for Baseline and Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Secukinumab Subcutaneous Injection
Number analyzed (Participants) | 4
score on a scale
  Week 1 | 1 (2)
  Week 24 | 1 (1.54)

4. Secondary Outcome: Dermatology Life Quality Index
Description: Number of subjects improving based upon patient-reported outcomes The Dermatology Life Quality Index (DLQI) is a validated general dermatology questionnaire that consists of 10 items that assess subject health-related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment)
  The scoring of each question is as follows:
  Very much scored = 3 points, A lot scored = 2 points, A little scored = 1, Not at all scored = 0 points, Not relevant scored = 0 points, Question 7, 'prevented work or studying' scored = 3 points. The DLQI is calculated by adding the score of each question, resulting in a maximum of 30 (meaning maximum impact on quality of life) and a minimum of 0 (meaning no impact of skin disease on quality of life). The higher the score, the more quality of life is impaired.
  0-1 = No effect on patient's life, 2-5 = Small effect, 6-10 = Moderate effect, 11-20 = Very large effect, 21-30 = Extremely large effect.
Time Frame: Baseline and Week 24
Population: DLQI data analyzed for Baseline and Week 24 only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Secukinumab Subcutaneous Injection
Number analyzed (Participants) | 4
score on a scale
  Week 1 | 6.25 (4.43)
  Week 24 | 3.25 (4.57)

ADVERSE EVENTS:
Time Frame: At every visit adverse events will be registered for 36 weeks
Description: Adverse events are defined as any undesirable experience occurring to a subject during the study, associated to the investigational treatment. All adverse events observed by investigator or staff members or reported by the subject will be recorded.
Arm/Group | Secukinumab Subcutaneous Injection
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT03791060/Prot_SAP_002.pdf
  • Informed Consent Form (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT03791060/ICF_005.pdf